CLINICAL TRIAL: NCT07145242
Title: Short-Term Effects of Acupuncture on Balance, and Quality of Life in Women With Migraine: A Pilot Study
Acronym: SAMBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Zaliene (Other)
Collaborators: Pain and Rehabilitation Medicine (Other)
Responsible Party: Sponsor-Investigator, Laura Zaliene, Lecturer, Klaipėda University, Klaipėda University
Organization: Klaipėda University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Approval No. 6 Sv-HMR-07
Record Dates: First submitted 2025-08-19; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Migraine
Keywords: acupuncture, migraine, medicine, balance, quality of life, pain mgmt, stress
MeSH Terms: conditions — Migraine Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short-Term Acupuncture for Migraine (Experimental): Participants in this arm received short-term acupuncture treatment specifically targeted for migraine accompanied by dizziness. The intervention consisted of six acupuncture sessions administered over a two-week period by a licensed acupuncturist. Standardized acupoints (GB7, GB14, GB20, GV20, LI4, LR3, Yintang) were used, with sterile disposable needles inserted according to traditional Chinese medicine guidelines. Each session lasted approximately 30 minutes. No comparator group was included, as this was a pilot exploratory trial.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Intervention Description * § Add details that will distinguish this intervention from other interventions in this or another clinical study.

SUMMARY:
The goal of this clinical trial is to learn about the short-term effects of acupuncture on migraine-related pain, postural balance, and quality of life in women with migraine.

The main questions it aims to answer are:

Does acupuncture reduce migraine pain intensity? Does acupuncture improve balance and postural stability in women with migraine? Does acupuncture improve quality of life in women with migraine? This study does not include a comparison group.

Participants will:

Receive six standardized acupuncture sessions over two weeks (three sessions per week).

Complete questionnaires on pain intensity (Visual Analogue Scale, VAS) and quality of life (SF-36).

Undergo stabilometric balance testing before and after the acupuncture program.

DETAILED DESCRIPTION:
Migraine is a highly prevalent neurological disorder characterized not only by recurrent headache attacks but also by associated symptoms such as dizziness, balance disturbances, and autonomic dysfunction. These vestibular comorbidities contribute to reduced functional capacity, higher risk of falls, and significantly diminished quality of life. Women of reproductive age are disproportionately affected, making this a critical population for targeted interventions. Conventional pharmacological treatments, while effective for some patients, are often associated with limitations including side effects, contraindications during pregnancy, and insufficient relief of vestibular symptoms. This underlines the need for safe, accessible, and integrative therapeutic approaches.

Acupuncture has gained increasing recognition as a complementary therapy for migraine. Previous clinical trials and meta-analyses have demonstrated its effectiveness in reducing headache frequency and intensity, as well as improving patient-reported quality of life. Proposed mechanisms include the modulation of central pain pathways, regulation of limbic and hypothalamic activity, activation of endogenous opioid release, and improvements in autonomic nervous system balance. However, relatively few studies have examined the effects of acupuncture on postural stability and vestibular-related outcomes in migraine populations, leaving a critical gap in the evidence base.

The current pilot clinical trial was designed to investigate the short-term effects of a standardized two-week acupuncture protocol on three domains:

Migraine pain intensity measured using a visual analogue scale (VAS). Postural stability assessed with stabilometric testing under eyes-open and eyes-closed conditions.

Health-related quality of life assessed with the SF-36 questionnaire. The study enrolled adult women with neurologist-confirmed migraine accompanied by dizziness. Eligible participants received six acupuncture sessions over two weeks, targeting acupoints traditionally linked with migraine relief and vestibular regulation (GB7, GB14, GB20, GV20, LI4, LR3, and Yintang). Treatment was delivered by a licensed acupuncturist, with strict adherence to protocol fidelity and safety monitoring.

The study was designed as a pilot randomized trial to evaluate feasibility and generate preliminary effect size estimates for future larger-scale studies. By focusing not only on pain but also on functional balance and quality of life, this trial expands the scope of acupuncture research in migraine and contributes novel data to an underexplored area.

The expected contribution of this trial is twofold: first, to provide early evidence on the multidimensional benefits of acupuncture in migraine with dizziness; and second, to inform the design, sample size calculation, and outcome selection for future randomized controlled trials. Given the non-invasive and low-risk nature of acupuncture, the findings may have particular clinical relevance for patients seeking integrative care approaches, including those with contraindications to pharmacological therapies.

ELIGIBILITY:
Inclusion criteria:

* Adult women (≥18 years)
* Neurologist-confirmed diagnosis of migraine according to the International Classification of Headache Disorders (ICHD-3)
* Presence of migraine-related symptoms, including recurrent headaches with or without aura
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Pregnancy
* Presence of other significant neurological or vestibular disorders
* Severe comorbidities that could interfere with balance assessment
* Contraindications for acupuncture treatment (e.g., skin infections at needling sites, bleeding disorders)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 12 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in migraine pain intensity measured by Visual Analogue Scale (VAS) | Baseline (Day 1) and at 2 weeks (end of intervention).
  Migraine pain intensity will be assessed using a 10 cm Visual Analogue Scale (VAS), where 0 indicates "no pain" and 10 indicates "worst imaginable pain." The primary outcome is the change in mean VAS score from baseline to 2 weeks post-intervention.

SECONDARY OUTCOMES:
Change in quality of life measured by SF-36 | Baseline (Day 1) and at 2 weeks (end of intervention)
  Quality of life will be assessed using the validated SF-36 Questionnaire, which evaluates the impact of migraine on daily functioning across role function, emotional function, and social domains. The secondary outcome is defined as the change in total MSQ score from baseline to 2 weeks post-intervention.
Change in postural balance measured by stabilometric platform | Baseline (Day 1) and at 2 weeks (end of intervention)
  Postural balance will be evaluated using a stabilometric platform by measuring center-of-pressure (COP) displacement in quiet standing. The outcome is defined as the change in mean sway path length and sway area from baseline to 2 weeks post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Zaliene, PhD, Principal Investigator — Klaipėda University
Locations (1):
- Klaipeda university, Klaipėda, Klaipėda County, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be shared due to the small sample size and the sensitive nature of health-related information. Ensuring participant privacy and compliance with ethical regulations precludes the public sharing of individual-level data.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT07145242/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT07145242/ICF_001.pdf